CLINICAL TRIAL: NCT06193005
Title: A Study of the Correlation Between Psychological Resilience and Genetic, Inflammatory Indicators in Young Population
Brief Title: Correlation Between Psychological Resilience and Genetic, Inflammatory Indicators
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Guang Zhang, Vice President, Qianfoshan Hospital
Other Study IDs: SDHMC-231202
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Genetic Predisposition to Disease; Environment; Adaptation, Psychological; Inflammation
MeSH Terms: conditions — Genetic Predisposition to Disease; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Form of biological specimen storage: venous blood was collected on an empty stomach, 5 ml was placed in a blood collection tube containing procoagulant and 5 ml was placed in a blood collection tube containing anticoagulant. Blood and other non-tissue samples are stored in a refrigerator at -86°C. The identification of the stored samples is unique and does not contain any donor identification information; the unique code is automatically and randomly generated by the sample bank management system and consists of 18 digits.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- very low adaptive group: The subjects were divided into very low adaptive group, low adaptive group, high adaptive group and very high adaptive group according to the quartile of adaptive ability score.
  Interventions: Other: no intervention
- low adaptive group: The subjects were divided into very low adaptive group, low adaptive group, high adaptive group and very high adaptive group according to the quartile of adaptive ability score.
  Interventions: Other: no intervention
- high adaptive group: The subjects were divided into very low adaptive group, low adaptive group, high adaptive group and very high adaptive group according to the quartile of adaptive ability score.
  Interventions: Other: no intervention
- very high adaptive group: The subjects were divided into very low adaptive group, low adaptive group, high adaptive group and very high adaptive group according to the quartile of adaptive ability score.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The goal of this observational study is to evaluate and analyze the influencing factors of the adaptive ability of young people, explore the impact of the interaction of environment and gene on the psychological adaptive ability of young people, incorporate the prediction model of the dynamic change of adaptive ability, build a standardized norm of young people's adaptive ability, and form a grading reference standard system. The main questions it aims to answer are:

* What are most important influencing factors for the adaptive ability of young people?
* How the environment and gene interact with each other on the psychological adaptive ability of young people?
* Can we build a prediction model of the dynamic change of adaptive ability and form a grading reference standard system?

Participants will support us with basic information data, adaptive ability assessment data, genetic testing data, brain image scanning data, and inflammatory indicators data. Then subjects were divided into very low adaptive group, low adaptive group, high adaptive group and very high adaptive group according to the quartile of adaptive ability score. And the statistical analysis will be performed by the data analyst.

DETAILED DESCRIPTION:
18-24 years old is an important stage of psychological development and personality shaping of young people. The higher cortex of the brain, which is responsible for emotional regulation and environmental coping, enters a critical period of neuroplasticity development. Its psychological development is characterized by transition, closure and turbulence, etc. When facing the stressful environment such as college entrance, employment and rapid social development, depression, anxiety and other negative emotional experiences may occur. All kinds of psychological problems. According to the critical period theory of emotional development, emotional states and stress coping are regulated by the activities of the brain's higher cortex. At the same time, the occurrence of mental disorders such as adaptation disorders is also influenced by genetics, and people with high-risk genes are more likely to have disorders.

The purpose of this study is to focus on the evaluation and analysis of the influencing factors of the adaptive ability of young people, explore the impact of the interaction of environment and gene on the psychological adaptive ability of young people, incorporate the prediction model of the dynamic change of adaptive ability, build a standardized norm of young people's adaptive ability, and form a grading reference standard system.

Research contents: 1) According to the cognitive theory system of adaptive ability and the individual prediction model of adaptive ability, considering the environmental characteristics that affect the adaptive ability of young people, the evaluation items with high predictive power of the model are screened. 2) Test the adaptive ability evaluation system in the research objects, verify the reliability, validity and extensibility of the task, and verify the measurement reliability and ecological validity of the paradigm tool. 3) Representative populations with high and low adaptive ability were selected to conduct multi-dimensional data collection on genetics and brain nerve, study the genetic risk and risk gene loci of adaptive ability, analyze the brain image features corresponding to adaptive ability, and study the neural mechanism of adaptive ability.

This study was designed as a cross-sectional study, with young people aged 18-22 as the research objects. The inclusion criteria included 18-22 years old, high school graduation or above, consent to blood sample collection, and signed informed consent. Exclusion criteria include not agreeing to take blood samples, not signing informed consent forms, and having a major medical condition such as a malignant tumor. It is planned to recruit 400 subjects from January 1, 2024 to March 31, 2024, and collect basic information data, adaptive ability assessment data, genetic testing data, brain image scanning data, and inflammatory indicators data.

The subjects were divided into very low adaptive group, low adaptive group, high adaptive group and very high adaptive group according to the quartile of adaptive ability score. A variety of predictive modeling techniques (such as Logistic discriminant model, neural network model, decision tree, random forest model and support vector machine, etc.) are used to construct a dynamic change prediction model adapted to outcome risk. The internal validation of the model was carried out by using the ten-fold cross-validation method. The original data were divided into 10 groups, among which 9 groups were taken as the training set and 1 group was taken as the test set for cross-validation to ensure the stability of the model. ROC curve was drawn to evaluate the differentiation of evaluation models. The area under ROC curve synthesizes two indexes of sensitivity and specificity, and considers every possible threshold value, which can evaluate the diagnostic value of the model more objectively and accurately. By calculating the area AUC under ROC curve as a quantitative analysis of the diagnostic value of the model, the closer the AUC is to 1, the better the diagnostic effect is. The Hosmer-Lemeshow goodness of fit test was used to judge the degree of consistency between the predicted risk and the actual risk, so as to evaluate the calibration degree of the model.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-24 years old; high school graduation and above; agree to collect blood samples and sign an informed consent form.

Exclusion Criteria:

* Did not consent to the collection of blood samples; did not sign an informed consent form; suffered from a major illness such as a malignant tumor.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 18-24 years old young people
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the Assessment of the Psychological Resillience | 1 year
  Psychological Resillience was evaluated across multiple dimensions, including cognitive functioning, stress coping, psychological well-being, and personality traits, and was measured using internationally accepted scales. Psychological Resillience is measured using the Psychological Resilience Scale (CD-RISC), which consists of 25 items rated on a 5-point Richter's scale, with scores ranging from 0 to 4 indicating that this is not the case at all, seldom the case, sometimes the case, often the case, and almost always the case. The sum of the scores of the items is the total score of the scale, and the total score is 0~100, the larger the score indicates the higher the level of psychological resilience, and the score of less than 60 is the poor level of psychological resilience, 61~69 is the average level of psychological resilience, 70~79 is the good level of psychological resilience, and >=80 is the excellent level of psychological resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Zhang, Dr, Principal Investigator — Qianfoshan Hospital

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Greenberg RL, Guzick AG, Schneider SC, Weinzimmer SA, Kook M, Perozo Garcia AB, Storch EA. Depressive Symptoms in Autistic Youth with Anxiety Disorders. J Dev Behav Pediatr. 2023 Dec 1;44(9):e597-e603. doi: 10.1097/DBP.0000000000001223. Epub 2023 Oct 11. PMID 38019467
- [Background] Brunette MF, Erlich MD, Edwards ML, Adler DA, Berlant J, Dixon L, First MB, Oslin DW, Siris SG, Talley RM. Addressing the Increasing Mental Health Distress and Mental Illness Among Young Adults in the United States. J Nerv Ment Dis. 2023 Dec 1;211(12):961-967. doi: 10.1097/NMD.0000000000001734. PMID 38015186
- [Background] Wong WLE, Arathimos R, Lewis CM, Young AH, Dawe GS. Investigating the role of the relaxin-3/RXFP3 system in neuropsychiatric disorders and metabolic phenotypes: A candidate gene approach. PLoS One. 2023 Nov 15;18(11):e0294045. doi: 10.1371/journal.pone.0294045. eCollection 2023. PMID 37967073